CLINICAL TRIAL: NCT01919541
Title: Understanding How Exercise and Nutrition Enhance Preoperative Functional Capacity: a Mechanistic Study
Brief Title: Mechanistic Prehabilitation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty in recruiting patients
Sponsor: Franco Carli (Other)
Responsible Party: Sponsor-Investigator, Franco Carli, Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 13-127-GEN
Record Dates: First submitted 2013-07-31; First posted 2013-08-09 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2015-09

CONDITIONS: Colon Cancer; Rectal Cancer
Keywords: Colorectal Surgery
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Preoperative Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Prehabilitation (Other): All patients will receive a prehabilitation program involving an individualized exercise and nutrition program 4 weeks before surgery. Whole body protein kinetics and insulin resistance will be determined at the beginning of the program and at the end of the program.
  Interventions: Other: Prehabilitation; Device: hyperinsulinemic euglycemic isoaminoacid clamp; Device: hyperinsulinemic euglycemic hyperaminoacid clamp; Dietary Supplement: whey protein supplementation

INTERVENTIONS:
Other: Prehabilitation — All patients will receive a prehabilitation program, which involves a personalized exercise component provided by a kinesiologist.
Device: hyperinsulinemic euglycemic isoaminoacid clamp — A hyperinsulinemic euglycemic isoaminoacid clamp followed by a hyperinsulinemic euglycemic hyperaminoacid clamp performed at baseline and immediately before surgery will provide insight into insulin resistance of glucose and protein metabolism in colorectal cancer patients pre- and post-intervention. Similarly, simultaneous infusions of leucine and glucose stable isotopes will provide insight into baseline and interventional effects of the program on whole body leucine and glucose kinetics.
Device: hyperinsulinemic euglycemic hyperaminoacid clamp
Dietary Supplement: whey protein supplementation
Other: Prehabilitation — All patients will receive nutrition guidance and a nutrition component with whey protein supplementation.

SUMMARY:
The investigators hypothesize that individuals who receive a personalized 4 week prehabilitation program consisting of exercise and nutrition counselling with post-workout whey protein supplementation will show, before colorectal surgery, improved insulin sensitivity, inflammatory profile, and substrate utilization compared to baseline measures. These results will translate into a higher functional capacity before surgery as demonstrated by an improvement in 6-minute walking test.

DETAILED DESCRIPTION:
Intervention Physical exercise program

At the baseline assessment all patients' physical fitness will be evaluated by the kinesiologist (exercise specialist). The exercise component will consist of approximately 60 min of resistance and aerobic training, for a minimum of 3 days per week. The exercise program will be individualized based upon the baseline fitness test (according to the American College of Sport Medicine, ACMS, standard)50 and will include: a 5 min warm-up, either 25 min of aerobic exercise (starting at 30- 40 % of heart rate reserve, HRR), and 25 min of resistance training (8 exercises targeting major muscle groups performed at moderate intensity), and a 5-10 min cool-down and stretching period. All exercises will be clearly explained and demonstrated by the kinesiologist at baseline. Patients will be asked to carry out this program at home, unsupervised, but will be monitored with weekly telephone calls. Training intensity progression will occur when the participant can complete aerobic exercise on mild exertion and/or when the participant can complete 15 repetitions of a given resistance exercise. Participants will be provided with resistance bands and an exercise mat, as well as a pedometer and a heart rate monitor, which can be used by the participant to monitor progress and by the kinesiologist to monitor daily compliance. A log book will also be completed to report all activities and frequency of exercises completed.

The kinesiologist will follow (by telephone call) all the participants on a weekly basis to ensure program compliance and address any barriers that may prevent ongoing participation.

Nutritional counseling The patients' nutritional status and adequacy of dietary intake will be assessed by a nutritionist using a three day food record, biological indices (e.g. glycated hemoglobin), clinical history, and the Patient-Generated Subjective Global Assessment tool51. Anthropometric measures, including percentage of lean body mass and fat, will be measured with bioelectrical impedance and skin calipers. Nutritional care plans will focus on meeting daily protein requirements (1.2g/kg), management of cancer-related symptoms (such as diarrhea, constipation), blood glucose control, optimization of body composition (i.e. weight loss/gain if necessary) and nutrient intake through providing practical suggestions, based on actual intake, to improve macronutrient distributions of protein, fat, and carbohydrates.

The type of dietary protein (amino acid composition), digestibility, amount, timing of intake, and co-ingestion with other macronutrients can be used to capitalize on post-exercise induced muscle protein synthesis52. Twenty (20) grams of protein, in liquid form, taken immediately after resistance exercise is regarded as sufficient to maximally stimulate muscle protein synthesis in healthy individuals52. Whey protein, in particular, is regarded as being especially effective when ingested after exercise54 because it is rapidly digested and contains all of the indispensable amino acids including leucine, which is believed to independently stimulate translation initiation of protein synthesis in skeletal muscle52. Post exercise co-ingestion with carbohydrate does not appear to provide any further anabolic effect, although does improve protein balance by blunting proteolysis and maximally stimulating insulin secretion55.

The nutritionist will provide patients with a post-workout nutrition prescription consisting of 20g of whey protein52 and 1g/kg carbohydrates53. Elderly patients require at least a 20g dose of dietary protein after resistance exercise and approximately 30g doses, in intervals, within the 24h "window of anabolic opportunity" in order to simulate an anabolic response 52.54,61. Ingestion of 1-1.5g carbohydrate/kg, within the "glycogen recovery window" of 15-30 minutes after exercise, replenishes glycogen stores53.

To ensure compliance, patients will be asked to complete daily logs and to return their empty sachets of whey protein.

Relaxation Strategies The kinesiologists will instruct patients to perform deep breathing exercises for relaxation purposes. Patients will be instructed to perform these exercises daily and as needed. Relaxation CD's, including soothing sounds, will also be given to patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective colorectal surgery for cancer
* 65 years and older

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) health status class 4-5
* disabling co-morbid physical and mental conditions (e.g. orthopedic and neuromuscular disease, dementia, psychosis)
* endocrine disorders (diabetes or hemoglobin A1C>6, hyper and hypothyrodisim)
* steroid consumption
* cardiac failure (New York Heart Association classes I-IV)
* chronic obstructive pulmonary disease
* renal failure (creatinine > 115µmol/l)
* hepatic failure (liver aminotranferases >50% the normal range)
* morbid obesity (BMI >40)
* anemia (hematocrit < 30 %, haemoglobin <100 g/L, albumin < 25 g/L)
* poor comprehension of English or French

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Protein Synthesis | up to 4 weeks before surgery
  The change in whole body protein synthesis, measured using stable isotope technology, from baseline to date of surgery, will be documented, in response to hyperinsulinemia with the use of a hyperinsulinemic euglycemic hyperaminoacidemic clamp.

CONTACTS AND LOCATIONS:
Overall Officials: Franco Carli, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Background] Li C, Carli F, Lee L, Charlebois P, Stein B, Liberman AS, Kaneva P, Augustin B, Wongyingsinn M, Gamsa A, Kim DJ, Vassiliou MC, Feldman LS. Impact of a trimodal prehabilitation program on functional recovery after colorectal cancer surgery: a pilot study. Surg Endosc. 2013 Apr;27(4):1072-82. doi: 10.1007/s00464-012-2560-5. Epub 2012 Oct 9. PMID 23052535
- See also: Related Info — http://www.mcgill.ca/peri-op-program/